CLINICAL TRIAL: NCT04780685
Title: A Phase II, Double-blind, Placebo-controlled Study to Assess the Safety, Tolerability, and Preliminary Efficacy of Intravenous Allogeneic Mesenchymal Stem Cells in Patients With Moderate to Severe ARDS Due to COVID-19
Brief Title: A Phase II Study in Patients With Moderate to Severe ARDS Due to COVID-19
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Stemedica Cell Technologies, Inc. (Industry)
Collaborators: bioRASI, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STEM-107-COVID-19
Record Dates: First submitted 2021-03-01; First posted 2021-03-03 (Actual); Last update posted 2022-07-08 (Actual); Status verified 2022-07

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is double-blind study
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- hMSCs (Experimental): hMSCs will be given via IV administration.
  Interventions: Biological: hMSC
- Lactated Ringer's Solution (Placebo Comparator): Lactated Ringer's Solution will be given via IV administration.
  Interventions: Biological: hMSC

INTERVENTIONS:
Biological: hMSC — IV administration
  Other Names: allogeneic mesenchymal bone marrow cells

SUMMARY:
This is a Phase II multi-center, double-blind, placebo-controlled, randomized study in Patients with moderate to severe lung injury due to COVID-19 or other potential viral and bacterial pathogens.

DETAILED DESCRIPTION:
This is a Phase II multi-center, double-blind, placebo-controlled, randomized study in Patients with moderate to severe lung injury due to COVID-19 or other potential viral and bacterial pathogens. The study will enroll up to 40 Patients into two cohorts, randomized 1:1 to receive active study drug plus standard treatment or placebo (LRS) plus standard treatment. On the treatment (Day 0) Cohort 1 will receive a single IV dose of hMSCs Cohort 2 will receive Lactated Ringer's Solution. A second dose of MSCs or LRS will be given to Cohort 1 or Cohort 2, respectively on Day 3 after the first dose. Patients who discontinue the study before Month 1 for reasons other than adverse events will be replaced.

ELIGIBILITY:
Inclusion Criteria:

* Laboratory-confirmed diagnosis of COVID-19 <= 14 days prior to randomization
* The presence of moderate to severe Acute Respiratory Distress Syndrome (ARDS) as defined by the Berlin Definition:

  1. Bilateral chest radiograph infiltrates.
  2. PaO2:FiO2 ratio of less than 200.
  3. Absence of other clinical conditions that could present in a similar manner (non-infectious pneumonitis, cardiogenic pulmonary edema)
* Absence of moribund state that would indicate imminent demise and poor chance of survival.

Exclusion Criteria:

* Females of childbearing potential who are pregnant or unwilling to undergo pregnancy testing; females with a positive pregnancy test on screening day will be excluded.
* Breastfeeding mothers
* Patients on ECMO
* Receiving concurrent treatment with an investigational agent in a clinical trial.
* Exception: Use of COVID-19 convalescent plasma is permitted.
* More than 72hrs on mechanical ventilation before randomization
* Receiving concurrent investigational vaccine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-03-20 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Survival | 14 days post treatment
  Number of patients alive at day 14 post treatment

SECONDARY OUTCOMES:
Number of patients with treatment-related adverse events as assessed by CTCAE v4.0 | 9 months
  Frequency of adverse events in patients treated with hMSCs and Lactate Ringer's solutions will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Lev Verkh, PhD/MS, Study Director — Stemedica Cell Technologies, Inc.; Santosh Kesari, MD, Principal Investigator — Providence Saint John's Health Center - Saint John's Cancer
Locations (2):
- United States (2):
  - Providence Medical Foundation, Fullerton, California
  - Providence Saint John's Health Center - Saint John's Cancer Institute, Santa Monica, California

IPD SHARING:
Plan to Share IPD: No